CLINICAL TRIAL: NCT03260023
Title: A Phase Ib/II Trial Evaluating the Combination of TG4001 and Avelumab in Patients With HPV-16 Positive Recurrent or Metastatic Malignancies.
Brief Title: Phase Ib/II of TG4001 and Avelumab in HPV16 Positive R/M Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); EMD Serono Research & Development Institute, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG4001.12
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HPV-Related Carcinoma; HPV-Related Cervical Carcinoma; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Penile Squamous Cell Carcinoma; HPV-Related Vulvar Squamous Cell Carcinoma
Keywords: Avelumab; Cancer; Anti PD-L1; Therapeutic Vaccine
MeSH Terms: conditions — Neoplasms | interventions — TG4001 vaccine; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TG4001/Avelumab (Experimental)
  Interventions: Biological: TG4001; Drug: Avelumab
- Avelumab (Experimental): Applicable for Phase II part 2.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Biological: TG4001 — PhIb: Dose escalation PhII: Established RP2D for TG4001
  Arms: TG4001/Avelumab
Drug: Avelumab — Anti PD-L1

SUMMARY:
The study will consist of two parts :

In the phase Ib: safety will be assessed in consecutive cohorts of 3 to 6 participants at increasing doses of TG4001 in combination with avelumab according to a 3+3 design. There will be no intra-participant dose escalation.

In the phase II part 1, evaluation of efficacy and further evaluation of safety of the combination of TG4001 and avelumab will be performed in a single arm of participants with recurrent or metastatic HPV-16 positive advanced malignancies.

In the phase II part 2, evaluation of efficacy of the combination of TG4001 and avelumab will be performed in a randomized, open-label controlled study comparing TG4001 in combination with avelumab to avelumab alone in participants with HPV-16 positive advanced malignancies.

In both phases, evaluation of tumor response will be done locally according to RECIST 1.1.

All participants will be followed up until disease progression, death, or unacceptable toxicity, or study withdrawal for any reason, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Female or male participants, aged at least 18 years (no upper limit of age)
* ECOG PS 0 or 1
* Life expectancy of at least 3 months
* Participants with histologically or cytologically documented metastatic or refractory/recurrent HPV-16 + cancer: cervical, vulvar, vaginal, penile and anal.
* Disease MUST not be amenable to curative surgery resection or curative radiotherapy with documented disease progression
* Prior therapy:

  * No more than one prior systemic treatment for recurrent /metastatic disease
  * Prior treatment for recurrent or metastatic disease is not required for:

    * Participants with recurrence/progression within 6 months after completion of prior multimodal therapy for localized or locally advanced disease
    * Participants who are unsuitable for platinum-based therapy
    * Participants who refuse chemotherapy or other standard therapies for the treatment of metastatic or recurrent disease
* Limited hepatic disease for participants with liver metastases at baseline
* Availability of tumor tissue from biopsy
* At least one measurable lesion by CT scan according to RECIST 1.1.
* Adequate hematological, hepatic and renal function
* Negative blood pregnancy test at screening for women of childbearing potential
* Highly effective contraception for both male and female participants if the risk of conception exists during the study period and for 3 months after the last study treatment administration

Exclusion Criteria:

* Prior exposure to cancer immunotherapy including cancer vaccines, any antibody/drug targeting T cell co-regulatory proteins (immune checkpoints)
* Participants under chronic treatment with systemic corticosteroids or other immunosuppressive drugs for a period of at least 4 weeks and whose treatment was not stopped 2 weeks prior to the first study treatment, with the exception of participants with adrenal insufficiency who may continue corticosteroids at physiological replacement dose, equivalent to ≤ 10 mg prednisone daily. Steroids with no or minimal systemic effect (topical, inhalation) are allowed
* Participants with CNS metastases except those with brain metastases treated locally and clinically stable during 4 weeks prior to start of study treatment, and those without ongoing neurological symptoms that are related to the brain localization of the disease
* Other active malignancy requiring concurrent systemic intervention
* Participants with previous malignancies other than the target malignancy to be investigated in this trial (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Participant with any organ transplantation, including allogeneic stem cell transplantation
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTC), any history of anaphylaxis, or uncontrolled asthma
* Any known allergy or reaction to eggs, gentamycin or attributed to compounds of similar chemical or biological composition to therapeutic vaccines/immunotherapeutic products
* Any known allergy or reaction to any component of anti-PD-L1/PD-1 or its excipients
* Participants with known history or any evidence of active interstitial lung disease / pneumonitis
* Participants with active, known, or suspected auto-immune disease or immunodeficiency, except type I diabetes mellitus, hypothyroidism only requiring hormone replacement or skin disorders (such as vitiligo, psoriasis) not requiring systemic treatment
* Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction (< 6 months prior to enrollment), unstable angina pectoris, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication/active intervention, history of myocarditis
* History of uncontrolled intercurrent illness including but not limited to:

  * Hypertension uncontrolled by standard therapies (not stabilized to 150/90 mmHg or lower)
  * Uncontrolled diabetes (e.g., hemoglobin A1c ≥ 8%)
  * Uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
- France (12):
  - I.C.O. Paul Papin, Angers
  - CHU Besançon, Besançon
  - Hôpital Saint André - CHU de Bordeaux, Bordeaux
  - Hôpitaux Civils de Colmar - Hôpital Pasteur, Colmar
  - CLCC Georges-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Curie, Paris
  - I.C.O. Gauducheau, Saint-Herblain
  - Centre Paul Strauss - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Institut Claudius Regaud - IUCT - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (6):
  - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Hospital Virgen de las Nieves, Granada
  - Fundación de Investigación biomédica H. 12 de Octubre, Madrid
  - Fundación de Investigación Biomédica Hospital Clínico San Carlos, Madrid
  - Hospital Virgen de La Victoria, Málaga
  - Hospital General de Valencia, Valencia

REFERENCES:
- [Result] Borcoman E, Lalanne A, Delord JP, Cassier PA, Rolland F, Salas S, Limacher JM, Capitain O, Lantz O, Ekwegbara C, Jeannot E, Cyrta J, Tran-Perennou C, Castel-Ajgal Z, Marret G, Piaggio E, Brandely M, Tavernaro A, Makhloufi H, Bendjama K, Le Tourneau C. Phase Ib/II trial of tipapkinogene sovacivec, a therapeutic human papillomavirus16-vaccine, in combination with avelumab in patients with advanced human papillomavirus16-positive cancers. Eur J Cancer. 2023 Sep;191:112981. doi: 10.1016/j.ejca.2023.112981. Epub 2023 Jul 11. PMID 37506588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 01 September 2017 through 27 March 2024, a total of 361 participants were screened.
  Phase Ib: 01 September 2017 until 11 April 2018 Phase II part 1: 04 October 2018 until 10 August 2020 Phase II part 2: 03 Jun 2021 until 27 March 2024
Pre-assignment Details: Out of 361 screened participants, 143 were included in the trial and 142 were administered with trial interventions. 218 participants were not included (main reasons: 48.6% inclusion criterion of having histologically or cytologically documented HPV-16+ cancer, 18.8% inclusion criterion of having adequate hematological, hepatic and renal function)
Groups:
- Phase I - TG4001 5x10e6 Pfu + Avelumab: Participants received 5x10e6 pfu TG4001 subcutaneously along with 10 mg/kg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase I - TG4001 5x10e7 Pfu + Avelumab; Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab: Participants received 5x10e7 pfu TG4001 subcutaneously along with 10 mg/kg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab; Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 Pfu + Avelumab: Participants received 5x10e7 pfu TG4001 subcutaneously along with 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab; Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab: Participants received 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Period: Overall Study
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab
Started | 3 | 6 | 34 | 46 | 44 | 5 | 5
Completed | 3 | 5 | 25 | 35 | 33 | 4 | 3
Not Completed | 0 | 1 | 9 | 11 | 11 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 4 | 4 | 4 | 1 | 2
Not completed — Clinical Progression | 0 | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Under trial intervention | 0 | 0 | 2 | 5 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In phase I and phase II part 1: all participants included and who received any amount of study treatment will be included in the SAF. Any participant who is assigned a participants number but does not receive any study treatment will not be included in the SAF.
  In phase II part 2: all randomized participants who were administered at least one dose of IMP(s) according to the treatment allocated at randomization will be included in the SAF.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab | Total
Number analyzed (Participants) | 3 | 6 | 34 | 46 | 44 | 5 | 4 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 25 | 37 | 30 | 4 | 2 | 104
  >=65 years | 0 | 3 | 9 | 9 | 14 | 1 | 2 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.0 [45.0 to 56.0] | 65.5 [51.0 to 68.0] | 56.0 [48.0 to 67.0] | 57.0 [50.0 to 61.0] | 56.5 [46.5 to 66.5] | 43.0 [41.0 to 54.0] | 67.5 [57.0 to 75.5] | 56.0 [48.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 25 | 43 | 44 | 5 | 4 | 125
  Male | 1 | 4 | 9 | 3 | 0 | 0 | 0 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  France | 3 | 6 | 34 | 39 | 37 | 4 | 4 | 127
  Spain | 0 | 0 | 0 | 6 | 7 | 1 | 0 | 14
Primary tumor location [Count of Participants; unit: Participants]
  Cervical | 0 | 1 | 8 | 25 | 24 | 3 | 0 | 61
  Anal | 2 | 0 | 17 | 14 | 13 | 2 | 4 | 52
  Oropharyngeal | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 10
  Vaginal | 0 | 1 | 3 | 2 | 3 | 0 | 0 | 9
  Vulvar | 0 | 0 | 1 | 4 | 4 | 0 | 0 | 9
  Penile | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Measure Description:
  The Eastern Cooperative Oncology Group (ECOG) score is an overall assessment of the functional/physical performance of the patient.
  Scores are:
  0=Fully active, able to carry on all pre-disease performance without restriction. 1=Restricted in strenuous activity but ambulatory and able to carry out work of a sedentary nature.
  Participants
    ECOG Status 0 | 0 | 4 | 10 | 18 | 11 | 3 | 1 | 47
    ECOG Status 1 | 3 | 2 | 24 | 28 | 33 | 2 | 3 | 95

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: To Evaluate the Safety and Tolerability of the Combination of TG4001 Plus Avelumab in Participants With Recurrent or Metastatic HPV-16 Positive Advanced Malignancies
Description: Dose limiting toxicities (DLTs) includes the following:
  * Grade ≥ 3 drug related adverse event (AEs). However, fatigue, nausea/vomiting adequately treated with anti-emetics, endocrinopathies adequately controlled with one physiologic hormone replacement, skin toxicity and single laboratory values out of normal range without any clinical correlate, asymptomatic grade ≥3 lipase or amylase elevation, tumor flare defined as local pain, irritation, or rash localized at sites of known or suspected tumor or a transient Grade 3 infusion adverse event are excluded.
  * Liver function test abnormality:
    * AST or ALT > 5 x ULN
    * Total bilirubin > 3 x ULN
    * Concurrent AST or ALT > 3 x ULN and total bilirubin > 2 x ULN
  * Drug related AE requiring treatment interruption for more than 2 weeks
Time Frame: From Day 1 to Day 28
Population: Phase Ib : All participants included and who received any amount of study treatment were included in the SAF. Any participant who was assigned a participant number, but did not receive any study treatment was not included in the SAF.
  Phase II part 1 and Phase II part 2: the outcome measure safety and tolerability has not been defined as primary endpoint.
  Therefore Phase II part 1 and Phase II part 2 are not included in the analysis population for safety and tolerability as primary endpoint.
Measure: Number; unit: DLT
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab
Number analyzed (Participants) | 3 | 6
DLT | 0 | 0

2. Primary Outcome: Phase II Part 1: Overall Response Rate (ORR) by RECIST 1.1
Description: Percentage of participants whose best overall response is either a Complete Response or a Partial Response according to Response Evaluation Criteria In Solid Tumors (RECIST v1.0) criteria over the the total number of evaluable participants.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: From treatment start, every 6 weeks for the first 9 months, then every 12 weeks up to 2 years.
Population: Phase II part 1 (Evaluable per protocol): Participants dosed with both IMPs and with at least baseline and post-baseline evaluable CT-scan at week 6 according to RECIST 1.1 and no major inc/exc, dosing or protocol violation, except if participant progressed or died due to disease.
  Phase Ib and phase II part 2: the outcome measure ORR has not been defined as primary endpoint.
  Therefore Phase Ib and phase II part 2 are not included in the analysis population for ORR as primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab
Number analyzed (Participants) | 30
percentage of participants
  Overall Response Rate | 16.67 [5.64 to 34.72]
  Disease Control Rate (DCR) | 46.67 [28.34 to 65.67]
  Complete Response (CR) | 3.33 [0.08 to 17.22]
  Partial Response (PR) | 13.33 [3.76 to 30.72]
  Stable Disease (SD) | 30.0 [14.73 to 49.40]
  Progressive disease (PD) | 53.33 [34.33 to 71.66]
Statistical Analysis 1: Comparison: Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab; A Simon's two-stage design will be used. The null hypothesis for response rate H0 is set at 10% corresponding to the response rate observed in second line participants, the alternate hypothesis of efficacy is set at HA=25%, the type I error α is set at 5% one sided, the type II error β is set at 20% (power=80%); Test type: Other — Enough participants will be treated to obtain 22 evaluable as a first stage. If at least 3/22 participants are considered responders, the enrolment will be continued, otherwise it will be stopped. For the second stage of the trial, enough participants will be treated to obtain a total of 40 evaluable participants and consider the study positive if at least 8/40 of them are considered responders; With a hierarchical strategy on the final analysis, a subgroup analysis performed in oropharyngeal SCCHN patients and with a null hypothesis for response rate (H0) set at 10% and the alternative hypothesis of efficacy set at HA = 35%, 18 oropharyngeal SCCHN patients would have been needed to reach a power of 81% and actual alpha at 2.8%. This analysis would have been considered positive with at least 5 responders among the 18 SCCHN patients. The second stage of the Simon's design has not been done following the decision to exclude oropharyngeal SCCHN and to change to a randomized controlled two-arms study (phase II part 2)

3. Primary Outcome: Phase II Part 2 Cohort A: Progression Free Survival (PFS) by RECIST 1.1
Description: PFS is defined as the time from the date of randomization to the date of first documented tumor progression or death due to any cause, whichever occurs first. If a participant has not had a PFS event at the cut-off date for analysis or at the date when a further antineoplastic therapy (other than those planned as study treatment in the protocol) is started, PFS will be censored at the date of last evaluable tumor assessment before the cut-off or start of further antineoplastic therapy.
Time Frame: From randomization: Every 6 weeks for the first 9 months, then every 12 weeks through study completion, for an average of 1 year.
Population: Phase II part 2, Cohort A: All randomized participants who were adminstered at least one dose of IMP(s) according to the treatment allocated at randomization. (FAS)
  For Phase Ib, Phase II part 1 and Phase II part 2 Cohort B : the outcome measure PFS has not been defined as primary endpoint Therefore Phase Ib, Phase II part 1 and Phase II part 2 Cohort B are not included in the analysis population for PFS as primary endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab: Participants without liver metastasis received 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Arm/Group | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab
Number analyzed (Participants) | 46 | 44
Months | 3.0 [2.0 to 4.4] | 2.8 [1.7 to 4.2]
Statistical Analysis 1: Comparison: Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab vs Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab; Efficacy will be evaluated by comparing the PFS between TG4001 arm versus TG4001 & avelumab arm with an adaptive approach. With one-sided type I error α at 5%, 76 events are needed to reach a power of 95%, corresponding to around 80 participants enrolled. To stick with initial timelines for final analyses and limiting the loss of statistical power, PFS analysis will be performed based on at least 69 events; Test type: Superiority — Statistical analysis is performed using a one-sided log-rank unstratified test to compare Progression-Free Survival of TG4001 in combination with avelumab vs avelumab alone in participants with recurrent or metastatic (R/M) HPV-16 positive advanced malignancies and without liver metastases at baseline. PFS will be evaluated based on RECIST1.1; p = 0.2810, Log Rank; Unstratified with one-sided p-value; Hazard Ratio (HR) = 0.87, 90% CI 2-sided [0.59 to 1.29]

4. Primary Outcome: Progression Free Survival (PFS) Phase II Part 2 Cohort A by Stratification
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Phase II part 2 Cohort A: All randomized participants who were adminstered at least one dose of IMP(s) according to the treatment allocated at randomization. (FAS)
  For Phase Ib, Phase II part 1 and Phase II part 2 Cohort B : the outcome measure PFS has not been defined as primary endpoint.
  Therefore Phase Ib, Phase II part 1 and Phase II part 2 Cohort B are not included in the analysis population for PFS as primary endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- Phase II Part 2 - Cohort A - Cervix Cancer - TG4001 5x10e7 Pfu + Avelumab; Phase II Part 2 - Cohort A - Anal Cancer - TG4001 5x10e7 Pfu + Avelumab; Phase II Part 2 - Cohort A - Genital Cancer - TG4001 5x10e7 Pfu + Avelumab: Participants without liver metastases received 5x10e7 pfu TG4001 subcutaneously along with 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase II Part 2 - Cohort A - Cervix Cancer - Avelumab; Phase II Part 2 - Cohort A - Anal Cancer - Avelumab; Phase II Part 2 - Cohort A - Genital Cancer - Avelumab: Participants without liver metastases received 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Arm/Group | Phase II Part 2 - Cohort A - Cervix Cancer - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Cervix Cancer - Avelumab | Phase II Part 2 - Cohort A - Anal Cancer - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Anal Cancer - Avelumab | Phase II Part 2 - Cohort A - Genital Cancer - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Genital Cancer - Avelumab
Number analyzed (Participants) | 25 | 24 | 14 | 13 | 7 | 7
Months | 4.3 [1.7 to 12.7] | 2.1 [1.4 to 2.8] | 3.0 [1.5 to 5.6] | 3.0 [1.4 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events. | 1.6 [1.4 to 5.6] | 7.2 [2.8 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events.

5. Secondary Outcome: Overall Response Rate (ORR) by Using RECIST 1.1 : Phase Ib, Phase II Part 2 Cohort A
Description: as for outcome 2
Time Frame: From treatment start (phase Ib) / randomization (phase II part 2) : Every 6 weeks for the first 9 months, then every 12 weeks up to 2 years.
Population: For Phase Ib / Phase II part 2 Cohort A: All participants who received at least one dose of IMP(s) according to treatment allocation.
  Phase II part 1 and phase II part 2 Cohort B: the outcome measure ORR has not been defined as secondary endpoint.
  Therefore Phase II part 1 and phase II part 2 Cohort B are not included in the analysis population for ORR as secondary endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab
Number analyzed (Participants) | 3 | 6 | 46 | 44
percentage of participants
  Overall Response Rate (ORR) | 0.0 | 50.0 | 15.2 | 13.6
  Disease Control Rate (DCR) | 33.3 | 83.3 | 65.2 | 68.2
  Complete Response (CR) | 0.0 | 0.0 | 8.7 | 2.3
  Partial Response (PR) | 0.0 | 50.0 | 6.5 | 11.4
  Stable Disease (SD) | 33.3 | 33.3 | 50.0 | 54.5
  Progressive Disease (PD) | 66.7 | 16.7 | 34.8 | 31.8
Statistical Analysis 1: Comparison: Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab vs Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab; In Phase II part 2 cohort A, statistical Test stratified by indication to compare the Overall Response Rate between TG4001+Avelumab versus Avelumab alone; Test type: Other; p = 0.832, Cochran-Mantel-Haenszel — At level 0.05 without adjustments for multiplicity testing, pvalue is calculated using Cochran-Mantel-Haenszel Chi-Square test

6. Secondary Outcome: Progression Free Survival (PFS) (Phase Ib, Phase II Part 1)
Description: PFS is defined as the time from the date of first study treatment administration (Phase Ib, Phase II Part1) to the date of first documented tumor progression or death due to any cause, whichever occurs first. If a participant has not had a PFS event at the cut-off date for analysis or at the date when a further antineoplastic therapy (other than those planned as study treatment in the protocol) is started, PFS will be censored at the date of last evaluable tumor assessment before the cut-off or start of further antineoplastic therapy.
Time Frame: From treatment start (phase Ib, phase II part 1): Every 6 weeks for the first 9 months, then every 12 weeks through study completion, for an average of 1 year.
Population: For Phase Ib: All participants included and who received any amount of study treatment.
  For phase II part 1: Evaluable participants population (EPP)
  Phase II part 2, cohort A and cohort B : the outcome measure PFS has not been defined as secondary endpoint.
  Therefore Phase II part 2, cohort A and cohort B are not included in the analysis population for PFS as secondary endpoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab
Number analyzed (Participants) | 3 | 6 | 30
Months | 1.6 [1.4 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events. | 12.0 [1.2 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events. | 1.5 [1.4 to 5.5]

7. Secondary Outcome: Overall Survival (OS) : Phase Ib, Phase II Part 1, Phase II Part 2 Cohort A
Description: Time from the date of first study treatment administration Phase Ib, Phase II part 1 or time from the date of randomization Phase II part 2 Cohort A to the date of death due to any cause.
  If a patient is not known to have died survival will be censored at the date of last contact.
Time Frame: From treatment start : Phase Ib, Phase II part 1 / from randomization: Phase II part 2 Cohort A through study completion, for an average of 4.5 years.
Population: Phase Ib: All participants included and who received any amount of study treatment.
  Phase II part 1: Evaluable participants' population. Phase II part 2 Cohort A: All randomized participants who were administered at least one dose of IMP(s) according to the treatment allocated at randomization.
  For the Phase II part 2 Cohort B, the outcome measure Overall Survival has not been defined as secondary endpoint. Therefore Phase II part 2 Cohort B is not included in the analysis population.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- Phase I - TG4001 5x10e6 Pfu: Participants received 5x10e6 pfu ofTG4001 subcutaneously along with 10 mg/kg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Arm/Group | Phase I - TG4001 5x10e6 Pfu | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab
Number analyzed (Participants) | 3 | 6 | 30 | 46 | 44
Months | 5.6 [5.6 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events. | 26.2 [8.7 to NA] — Upper limit of Confidence Interval has not been achieved due to insufficient number of participants with events. | 10.3 [6.2 to 13.3] | 16.6 [10.5 to 21.7] | 16.5 [10.0 to 19.6]

8. Secondary Outcome: Duration of Overall Response (DoR): Phase Ib, Phase II Part 1, Phase II Part 2 Cohort A
Description: Duration of overall response in weeks (DoR) applies only to patients whose best overall response is CR or PR. The start date is the date of first documented response (CR or PR) and the end date is the date of event defined as first documented disease progression or death due to underlying cancer.
Time Frame: From treatment start Phase Ib, Phase II part 1 / from randomization Phase II part 2 Cohort A : every 6 weeks for the first 9 months, then every 12 weeks through study completion, for an average of 2.5 years.
Population: For phase Ib, phase II part 1 and phase II part 2 Cohort A, analysis population consists of all included participants who were dosed with IMP(s) according to treatment allocation and who have a confirmed response according to RECIST1.1.
  For Phase II part 2 Cohort B, the outcome measure duration of overall response has not been defined as secondary endpoint. Therefore Phase II part 2 cohort B is not included in the analysis population.
Measure: Median (Full Range); unit: Weeks
Groups:
- Phase I - TG4001 5x10e6 Pfu Avelumab: Participants received 5x10e6 pfu TG4001 subcutaneously along with 10 mg/kg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase I - TG4001 5x10e7 Pfu Avelumab; Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab: Participants received 5x10e7 pfu TG4001 subcutaneously along with 10 mg/kg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Arm/Group | Phase I - TG4001 5x10e6 Pfu Avelumab | Phase I - TG4001 5x10e7 Pfu Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab
Number analyzed (Participants) | 0 | 3 | 5 | 7 | 6
Weeks |  | 53.7 [40.7 to 239.7] | 25.1 [22.4 to 228.1] | 90.3 [12.1 to 138.4] | 55.9 [18.3 to 121.0]

9. Secondary Outcome: Proportion of Progressive Disease Phase II Part 2 Cohort B
Description: Number of participants with liver metastases at baseline who has a documented disease progression as per RECIST1.1.
Time Frame: From randomization: every 6 weeks up to 24 weeks.
Population: Phase II part 2 Cohort B: All randomized participants administered with at least one dose of IMP(s) according to allocation at randomization (FAS). One participant (cohort B - Avelumab) was excluded from analysis because no IMP has been administered.
  Phase Ib, Phase II part 1 and Phase II part 2 Cohort A, proportion of progressive disease has not been defined as secondary endpoint. Therefore phase Ib, Phase II part 1 and Phase II part 2 Cohort A are not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab
Number analyzed (Participants) | 5 | 4
Participants
  Non progressive disease | 2 | 0
  Progressive disease <= 6 weeks | 2 | 1
  Progressive disease <= 12 weeks | 3 | 3
  Progressive disease <= 24 weeks | 3 | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed for up to 4.5 years. All non serious AEs not treatment related were reported from start of study treatment up to 30 days after last administration of study treatments through study completion for an average of 7 months. All treatment related non serious AEs and all SAEs were reported from start of study treatment up to 90 days after last administration of study treamtents through study completion for an average of 8.5 months.
Groups:
- Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab: Participants without liver metastasis received 5x10e7 pfu TG4001 subcutaneously along with 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
- Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 PFU + Avelumab: Participants with liver metastasis received 5x10e7 pfu TG4001 subcutaneously along with 800 mg avelumab intravenously until disease progression, unacceptable toxicity, participant withdrawal from study for any reason.
Arm/Group | Phase I - TG4001 5x10e6 Pfu + Avelumab | Phase I - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 PFU + Avelumab | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/6 | 12/34 | 7/46 | 5/44 | 1/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/6 | 18/34 | 16/46 | 18/44 | 2/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 34/34 | 46/46 | 43/44 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - TG4001 5x10e6 Pfu + Avelumab (N=3) | Phase I - TG4001 5x10e7 Pfu + Avelumab (N=6) | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab (N=34) | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab (N=46) | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab (N=44) | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 PFU + Avelumab (N=5) | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Central nervous system vasculitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - TG4001 5x10e6 Pfu + Avelumab (N=3) | Phase I - TG4001 5x10e7 Pfu + Avelumab (N=6) | Phase II Part 1 - TG4001 5x10e7 Pfu + Avelumab (N=34) | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - TG4001 5x10e7 Pfu + Avelumab (N=46) | Phase II Part 2 - Cohort A - Participants Without Liver Metastases - Avelumab (N=44) | Phase II Part 2 - Cohort B - Participants With Liver Metastases - TG4001 5x10e7 PFU + Avelumab (N=5) | Phase II Part 2 - Cohort B - Participants With Liver Metastases - Avelumab (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 15 (26) | 17 (43) | 13 (29) | 2 (4) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (4) | 5 (15) | 3 (7) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (12) | 2 (2) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (4)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 4 (4) | 8 (8) | 5 (5) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 3 (4) | 7 (7) | 3 (4) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 9 (10) | 8 (13) | 1 (2) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 13 (14) | 9 (12) | 10 (18) | 1 (1) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (6) | 5 (12) | 17 (23) | 13 (28) | 4 (6) | 2 (11)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malignant dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (9) | 8 (9) | 6 (10) | 1 (1) | 2 (6)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7) | 9 (14) | 6 (8) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (4) | 9 (14) | 16 (29) | 14 (27) | 1 (1) | 2 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 4 (4) | 10 (11) | 5 (8) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 8 (11) | 9 (17) | 10 (22) | 2 (5) | 2 (5)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 4 (6) | 8 (16) | 12 (29) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (15) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 5 (11) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 2 (4) | 5 (15) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 6 (7) | 8 (15) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 7 (8) | 8 (12) | 0 (0) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Medical device site joint pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 6 (7) | 7 (11) | 5 (11) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (6) | 3 (6) | 14 (25) | 18 (37) | 8 (13) | 2 (3) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 2 (2) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Cystitis escherichia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (4) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Root canal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 10 (15) | 2 (2) | 3 (3) | 2 (3) | 0 (0)
Vaginal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 4 (6) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 5 (6) | 5 (7) | 2 (2) | 1 (1) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal transit time increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (4) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 11 (12) | 11 (11) | 3 (4) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (8) | 2 (3) | 4 (6) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 6 (7) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (5) | 4 (4) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypozincaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (9) | 11 (19) | 9 (16) | 2 (3) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (4) | 8 (10) | 8 (13) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (11) | 3 (3) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 4 (5) | 1 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 10 (15) | 9 (12) | 8 (13) | 1 (1) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 8 (18) | 6 (12) | 1 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resting tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (7) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 3 (6) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 3 (3) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Ureteral spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine cervical pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 9 (10) | 6 (7) | 1 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 7 (7) | 4 (7) | 3 (3) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal reflux (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery occlusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 4 (4) | 6 (10) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (6) | 0 (0) | 0 (0)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Lymphostasis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03260023/Prot_SAP_002.pdf